CLINICAL TRIAL: NCT00073684
Title: Young Sexually Abused Children: Optimal CBT Strategies
Brief Title: Optimal Treatment Strategies for Sexually Abused Children
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rowan University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH064776 (NIH); R01MH064776 (NIH); DSIR 84-CTS
Record Dates: First submitted 2003-12-02; First posted 2003-12-03 (Estimated); Last update posted 2014-05-08 (Estimated); Status verified 2014-05

CONDITIONS: Child Abuse, Sexual
Keywords: Stress Disorders, Post-Traumatic; Depression; Anxiety
MeSH Terms: conditions — Coitus; Stress Disorders, Post-Traumatic; Depression; Anxiety Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- 1 (Experimental): Participants will receive 8 sessions of TF-CBT with narrative.
  Interventions: Behavioral: Trauma focused cognitive behavioral therapy (TF-CBT); Behavioral: Brief abuse-focused treatment
- 2 (Experimental): Participants will receive 8 sessions of TF-CBT without narrative.
  Interventions: Behavioral: Trauma focused cognitive behavioral therapy (TF-CBT); Behavioral: Brief coping skills treatment
- 3 (Experimental): Participants will receive 16 sessions of TF-CBT with narrative.
  Interventions: Behavioral: Trauma focused cognitive behavioral therapy (TF-CBT); Behavioral: Extended abuse-focused treatment
- 4 (Experimental): Participants will receive 16 sessions of TF-CBT without narrative.
  Interventions: Behavioral: Trauma focused cognitive behavioral therapy (TF-CBT); Behavioral: Extended coping skills treatment

INTERVENTIONS:
Behavioral: Trauma focused cognitive behavioral therapy (TF-CBT) — This study aims to: (1) examine the differential effects of CBT with and without trauma narrative interventions; (2) examine the comparative efficacy of brief and extended (8 vs. 16 sessions) individual CBT; (3) make developmental comparisons between 4-7 year olds and 8-11 year olds as to the appropriateness and therapeutic necessity of exposure interventions and longer treatment; and (4) identify child and parent factors that may significantly mediate the relationships between treatment conditions and outcomes. The findings of this study will help establish clinical as well as developmental markers for the early identification of sexually abused children who may require more focused (i.e., including trauma narrative) and/or longer treatment to achieve optimal outcomes.
Behavioral: Brief abuse-focused treatment — Participants will receive 8 sessions of TF-CBT with abuse-focused treatment.
  Arms: 1
Behavioral: Brief coping skills treatment — Participants will receive 8 sessions of TF-CBT with brief coping skills treatment.
  Arms: 2
Behavioral: Extended abuse-focused treatment — Participants will receive 16 sessions of TF-CBT with extended abuse-focused treatment.
  Arms: 3
Behavioral: Extended coping skills treatment — Participants will receive 16 sessions of TF-CBT with extended coping skills treatment.
  Arms: 4

SUMMARY:
This study will determine the necessity of including abuse-focused interventions in the treatment of sexually abused children.

DETAILED DESCRIPTION:
Child sexual abuse is a serious public health problem that places children at high risk for developing anxiety, mood, conduct, sexual, and substance abuse disorders. It also increases their likelihood of experiencing further victimization. It is imperative that abused children are provided with effective interventions to minimize their risk of developing problems that can be disruptive to their psychosocial development. Evidence suggests that cognitive behavioral therapy (CBT) can effectively ameliorate many abuse-related symptoms exhibited by sexually abused children and their parents. However, it is unknown whether CBT treatment should include gradual exposure (GE), an intervention that involves the gradual confrontation of abuse-related thoughts and memories with therapist feedback to assist the child in effectively processing the abusive experience. Because this component of CBT may be more difficult for children and their parents, it is important to determine if and when GE is essential for optimal recovery in abused children.

Children and their parents will be randomly assigned to receive one of four treatments: brief abuse-focused treatment, brief coping skills treatment, extended abuse-focused treatment, and extended coping skills treatment. Assessments will be conducted before, during, and after treatment and at 6- and 12-month follow-up visits. Standardized evaluations will be conducted to assess parents' distress and support levels; parent reports of children's behavior patterns, sexualized behaviors, and post-traumatic stress disorder (PTSD) symptoms; and children's self-reports of PTSD, depression and anxiety symptoms, body safety skills, and victimization experiences.

ELIGIBILITY:
Inclusion Criteria:

* Sexual abuse that has occurred within 24 months of the study. The abuse must have been substantiated by child protective services, charges must have been pressed by the prosecutor's office, or there must have been independent confirmation of abuse by a professional with recognized expertise in conducting investigative evaluations.
* Kiddie-Sads-Present and Lifetime Version (K-SADS-PL) criteria for partial or full post-traumatic stress disorder (PTSD)
* Parental consent
* Caretaker who has not abused the child

Exclusion Criteria:

* Mental Retardation (IQ less than 70) or placement in special education classes
* DSM-IV criteria for Pervasive Developmental Disorders
* Psychotic disorder
* Serious medical illness that could interfere with the study
* In temporary, emergency foster care. If a child is returned home or placed in short-term foster care that is anticipated to last a minimum of 4 months, then the child is eligible for participation.
* Parent who meets DSM-IV criteria for a psychotic disorder
* Parents with serious mental health problems that result in substantial functional impairment
* Unsupervised contact with abuse perpetrator
* Receiving concurrent psychiatric treatment for the abuse. If participants previously received sexual abuse treatment that did not resolve symptomology, they are eligible to participate. In addition, children who have contact with a psychiatrist for medication monitoring purposes may be included if their medication and dosage have remained stable for at least 6 weeks prior to study start

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 210 (Actual)
Dates: Start 2003-08; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
K-SADS-PL PTSD | Measured at Months 6 and 12

SECONDARY OUTCOMES:
Child Depression Inventory (CDI) | Measured at Months 6 and 12

CONTACTS AND LOCATIONS:
Locations (1):
- CARES Institute, Stratford, New Jersey, United States